CLINICAL TRIAL: NCT07293741
Title: The Impact of Virtual Doula Services on Birth Outcomes in Rural Communities
Acronym: RIVER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Lori Uscher-Pines, Senior Policy Researcher, RAND
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2R01NR018837-06 (NIH); 2R01NR018837-06 (NIH)
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Birth; Telehealth; Pregnancy; Maternal Health
Keywords: telehealth; virtual; doula; pregnancy; birth; maternal health

STUDY DESIGN:
Intervention Model Description: 2-arm, parallel design
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator Arm (Active Comparator): This arm will receive a free ebook on parenting. The care that they receive for pregnancy and birth will be care as usual.
  Interventions: Other: Ebook
- Virtual Doula Support (Experimental): This arm will receive up to 4 scheduled visits with doulas via a mobile phone app. Visits can be used any time throughout the perinatal period, including postpartum.
  Interventions: Other: Virtual doula support

INTERVENTIONS:
Other: Virtual doula support — Participants randomized to the intervention arm will receive access to up to 4 scheduled doula visits through Pacify's mobile phone app. All visits will be virtual. Participants may also access the library of resources on the app and text with their doula on demand.
  Arms: Virtual Doula Support
Other: Ebook — Participants will receive an ebook on parenting.
  Arms: Active Comparator Arm

SUMMARY:
This study will assess the impact of virtual doula care on birth and postnatal outcomes among rural mothers. The goal of virtual doula services is to improve access to care in underserved communities and decrease urban-rural differences in key maternal health outcomes including mode of birth (cesarean vs vaginal) and birth satisfaction. By implementing a digital randomized controlled trial, the study team will efficiently recruit a national sample of rural pregnant women to provide evidence of the effectiveness of virtual doula care, the appropriateness of virtual visits for different care and support needs, and the role of virtual care in improving maternal health.

DETAILED DESCRIPTION:
Rates of maternal morbidity have been rising in the U.S., and there are stark rural-urban differences in cesarean births and adverse pregnancy outcomes. Increasing access to doula care is a promising strategy to improve maternal health. Doulas are non-clinical providers who offer physical, emotional, and informational support throughout the perinatal period. Yet, despite documented evidence of effectiveness, fewer than 10% of U.S. births involve doulas because of costs and workforce shortages. Virtual doula services may increase access to support in communities that lack doulas and decrease costs; however, there is minimal evidence of the effectiveness of this new care model. Lack of research in general, and randomized controlled trials in particular, represents a significant gap given that virtual doula services are currently offered by numerous organizations, and the states and payers adding doula benefits do not have evidence to inform their telehealth policies.

The study team will conduct an innovative digital, parallel design randomized controlled trial (RCT) to assess the impact of virtual doula services in rural communities. Primiparous, pregnant women who live in rural zip codes in the U.S. will be recruited. Recruitment will occur via online research panels. Participants will be randomized to scheduled visits with virtual doulas throughout the perinatal period or to usual care. Birth and postnatal outcomes will be captured via surveys and interviews. This study uses mixed methods and aims to assess the impact of virtual doula services on primary outcomes including type of birth (cesarean vs vaginal), birth satisfaction, and parental self-efficacy and secondary outcomes including maternal depression, breastfeeding initiation and duration, and receipt of prenatal and postnatal care. This study will also explore the acceptability of virtual care for different types of doula visits. Together, these aims will inform policy debates about regulation and reimbursement of doula services that incorporate virtual care.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* pregnant (second or early third trimester) with their first child
* reside in a rural zip codes in the U.S.

Exclusion Criteria:

* non-singleton pregnancy
* police custody or incarceration
* infant to be separated from mother (e.g., placed for adoption, protective custody)
* working with a doula prior to enrollment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 614 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Birth type | Assessed at 3 weeks postpartum
  Cesarean or Vaginal Birth
Birth Satisfaction | Assessed at 3 weeks postpartum
  Score on Birth Satisfaction Scale-Revised. Scores can range from 0-40, with higher scores indicating greater satisfaction.
Parental Self-Efficacy | Assessed at 12 weeks postpartum
  Score on maternal confidence questionnaire. Scores can range from 14 to 70, with higher scores indicating greater maternal confidence.

SECONDARY OUTCOMES:
Maternal Depression | Assessed at 3 weeks postpartum
  Score on Edinburgh Depression Scale. Minimum score of 0 and maximum score of 27, with higher scores indicating increased severity of depressive symptoms.
Breastfeeding duration | Assessed at 12 weeks postpartum
  Any breastfeeding (yes/no) in prior 7 days
Receipt of postnatal care | Assessed at 12 weeks postpartum
  Attendance at postpartum visit
Birth Truma | Assessed at 3 weeks postpartum
  Traumatic birth experience (yes/no)
Breastfeeding Initiation | Assessed at 12 weeks postpartum
  Attempted breastfeeding (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- RAND, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide de-identified patient-level survey data on all primary and and secondary outcomes as well as demographic data. Data will be available in CSV format on the Harvard Data Respository
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available one year after the completion of the project and will be available for 5 years.
Access Criteria: Access to the scientific data will be made available by the Harvard Data Repository after a request has been submitted and approved by the PIs. To be approved, the requesting organization or individual should demonstrate that they intend to use the data for research purposes and that they have obtained IRB approval.
URL: https://dataverse.harvard.edu/